# Examining the Effectiveness of Cognitive Training

NCT04344028

4/30/2024

**Title of the Study:** Examining the Effectiveness of Cognitive Training

Principal Investigator: C. Shawn Green

Phone: (608) 263-4868; email: csgreen2@wisc.edu

## **DESCRIPTION OF THE RESEARCH**

You are invited to participate in a research study about how training can impact performance on cognitive tasks. You have been asked to participate because you are an adult 18 years of age or older, have normal (or corrected to normal) vision, and have no neurological conditions that would preclude your ability to complete computerized cognitive tasks. This research will take place in the laboratory of Dr. C. Shawn Green in the Department of Psychology at the University of Wisconsin-Madison.

## WHAT WILL MY PARTICIPATION INVOLVE?

If you decide to participate in this research you will first complete two sessions (~75 minutes each) where you are asked to view visual stimuli (such as black and white lines, letters, simple shapes like triangles, circles, and squares) presented on a computer or television screen and/or listen to auditory stimuli (such as pure tones) presented via headphone or speakers. You will then be asked to make some simple judgments about the stimuli (such as indicating whether the stimulus you observed is the same or different from that on a previous trial), and indicate your judgment decision with a button press on a keyboard, a mouse click, or a movement on a touchpad. You will also be asked to complete a set of questionnaires (please note you can skip any questions you are not comfortable answering).

After these initial sessions you may or may not be asked to complete two sets of 10 sessions (~20 minutes) of cognitive tasks either at home or in the lab. Each set of sessions should be completed over a period of no more than 15 days. If you are asked to do these sessions, you will be given instructions regarding the tasks you need to complete in these training sessions (which will be similar to some of the tasks you complete in the first two sessions, ~20 minutes) prior to these sessions. Should you be asked to complete those sessions at home, you will be provided a tablet to take home with you. The research group may contact you over this period to ensure you remain on schedule.

After completing the first set of 10 sessions, you will then return to the lab to complete one session (~75 minutes) of tasks similar to those you complete in the first sessions. If you were not asked to complete the 20-minute sessions, then you will come back to the lab about two weeks after the first two 75-minute sessions.

After you have completed this 75-minute session, you will be asked to come back to the lab after you have completed your second set of 20-minute sessions, or about a period of two weeks if you are not asked to complete the 20-minute sessions of cognitive tasks. Finally, after a couple of weeks, you will come back for your two final testing sessions (~45 minutes each). If you were provided with a tablet, you will also return it during the last session.

The total duration of the study will be around 8 hours if you are not asked to do the twenty 20-minute sessions, or 15 hours if you are asked to complete these sessions. The whole experiment runs over the course of 4 to 8 weeks. If you have questions about the time commitment, please inform the experimenter now.

#### ARE THERE ANY RISKS TO ME?

There are no major risks. Some of the tasks may induce a sense of boredom or fatigue. Please remember that you may interrupt or terminate your participation for any reason, including discomfort, and can do so at any time. There is always a small risk of a breach of confidentiality. However, all care will be taken to ensure that your data cannot be linked to your name.

#### ARE THERE ANY BENEFITS TO ME?

There are no direct benefits to participation.

## WILL I BE COMPENSATED FOR MY PARTICIPATION?

Depending on the group to which you are assigned to complete, you will receive either \$100 if you are assigned to the testing only group [7 in-lab sessions, 8 hours total], or \$200 if you are assigned to the training group [9 in-lab sessions + 20 in-lab or at-home sessions, 15 hours total] if you complete all the aspects of the study within the allowed timeframe. The experimenter will have discussed exact details of payment prior to your being given this form. If you do withdraw prior to the end of the study, you will receive compensation for the time that you completed prior to withdrawing from the study at a rate of \$10/hr.

#### HOW WILL MY CONFIDENTIALITY BE PROTECTED?

While there will probably be publications as a result of this study, your name will not be used. This study involves a collaboration between researchers at three sites – the University of Wisconsin-Madison, the Northeastern University (Boston, MA), and the University of California-Riverside. Data will be shared across all three sites, however, information about identity will not be shared with other sites (i.e., data will utilize a unique code and the link between that code and identity will be not be shared across sites). Furthermore, completely de-identified data may be shared with other researchers for future research without additional consent (i.e., the data will be put into a format where it will be impossible to identify you). Research data will be stored on a secure server separately from any identifying information, which will be kept in a secured area in locked room in the PIs lab space (for physical records) or in a password-protected file on a secure server. Finally, a description of this research study will be available on www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time. If you participate in this study, we would like to be able to quote you directly without using your name. If you agree to allow us to quote you in publications, please initial the statement at the bottom of this form.

If you sign this document, you give permission to the research team at UW-Madison to use or disclose (release) research records. This information may only be used by and/or disclosed (released) to representatives of the National Institute on Aging, the funding agency, and its authorized representatives, as well as representatives of UW-Madison's IRB (Institutional Review Board).

## WHOM SHOULD I CONTACT IF I HAVE QUESTIONS?

You may ask any questions about the research at any time. If you have questions about the research after you leave today you should contact the Principal Investigator, Christopher Shawn Green at (608) 263-4868.

For more information about participation in a research study and about the Institutional Review Board (IRB), your rights as a research participant, or if you have complaints about the research study or study team, please call the confidential research compliance line at 1-833-652-2506. Staff will work with you to address concerns about research participation and assist in resolving problems.

Your participation is completely voluntary. If you decide not to participate or to withdraw from the study, you may do so without penalty or, if applicable, effect on your grade. Your signature indicates that you have read this consent form, had an opportunity to ask any questions about your participation in this research and voluntarily consent to participate. You will receive a copy of this form for your records.

## WHO IS FUNDING THIS STUDY?

This study is funded by the NIA Grant Ro1-MSN251937awarded to C. Shawn Green, Aaron R. Seitz, and Susanne M. Jaeggi.

### PARTICIPANT SIGNATURE

By signing this consent form, you indicate that you discussed this study with an experimenter, reviewed the information in this form, had the opportunity to ask and appropriately answered any questions you may have, and are voluntarily choosing to take part in this research.

| Name of Participant (please print): | |
|---|---|
| Signature: | Date: |
| I give my permission to be quoted directly (initial): | in publications without using my name |
| I <u>would</u> / <u>would not</u> be interested in being (circle one above) | contacted to participate in future research. |
| EXPERIMENTER SIGNATURE | |
| Your signature below means that you have have answered any questions they have abo | explained the research to the participant and out the research. |
| Name of experimenter (Please Print) : | |
| Signature: | Date: |